CLINICAL TRIAL: NCT06086093
Title: Evaluate the Efficacy of RespireAidTM in Patient With Externally Contracted Seasonal Epidemic (外感時疫)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Ten Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MOHW-112-CM3B-01
Record Dates: First submitted 2023-10-03; First posted 2023-10-17 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Respiration Disorders
Keywords: RespireAid; Externally Contracted Seasonal Epidemic
MeSH Terms: conditions — Respiration Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo (Placebo Comparator): Take 1 sachet(5g) 4 times daily.
  Interventions: Dietary Supplement: RespireAid TM/placebo
- RespireAid (Experimental): Take 1 sachet(5g) 4 times daily.
  Interventions: Dietary Supplement: RespireAid TM/placebo

INTERVENTIONS:
Dietary Supplement: RespireAid TM/placebo — Direction: Take 1 sachet(5g) 4 times daily
  Indication: Externally contracted seasonal epidemic
  Function: Relieving Exterior and Facilitating Lung, clear heat of lung, Wide chest and resolve phlegm

SUMMARY:
The goal of this clinical trial is to learn about in the main objective of this study is to evaluate the clinical efficacy of the RespireAidTM (Tai-wan-Qing-Guan-Yi-Hao) to ease the symptoms of fever, sore throat, and cough, and the safety after treatment. Participants will Take 1 sachet(5g) 4 times daily. There is a comparison group: Researchers will compare placebo to see if RespireAidTM.

DETAILED DESCRIPTION:
This is a multicenter, parallel, double-blind, randomized, placebo-controlled study. A total of 258 male or unpregnant female outpatient subjects ≥ 18 years to ≤ 79 years of age will be enrolled into this study (dropout rate 10%). There will be 2 visits in this study. In Visit 1 (Day 1), subjects who have the symptoms of fever, sore throat, and cough (match the definition in table 1 to 3 in protocol), by investigator's judgement will be recruited into the study. Subjects will be randomized into the RespireAidTM group or placebo group with allocation rate 2:1. Following to the clinical guideline of NRICM101, subjects in RespireAidTM group will take drug four times daily with 20g oral granule, administered for 5 days. The subjects in placebo group received study drug with the same dose frequency. Other than study drugs, the rescue drug, acetaminophen, will be administered. If subjects have moderate or severe fever, sore throat, he/she could receive one rescue medication (500mg) per 4 hours, up to 6 tablets in total in one day. Subjects will be educated how to use e-dairy. The dairy will be recorded the severity of fever, sore throat, and cough from baseline (Day 1, before use of study drug) to Day 5. The efficacy endpoint will be the improvement of fever, sore throat, and cough, and the safety endpoint will be adverse events after treatment. The study and rescue drugs will be dispensed to subjects and the study staff will teach them how to receive medications. If subjects have persistent fever, unscheduled visits will be arranged to check whether or not they would be suitable to participate into this study.

Adverse events will be recorded at Visit 2(Day 8), and the dairy with drug record will be checked.

ELIGIBILITY:
Inclusion Criteria:

1. Male or unpregnant female patients ≥ 18 years to ≤ 79 years of age, who have the symptoms of fever, sore throat, and cough (match the definition in table 1 to 2 in protocol), by investigator's judgement, with mild to severe symptoms (> 20 mm in each VAS).
2. With BMI between 18 to 30 kg/m².
3. Without a history for alcohol or drug abuse, or other significant organic diseases.
4. No history of cancer. Unless no signs of relapse occurred for over 5 years which no anticancer therapies are needed.
5. Ability to read and write Chinese, and provide data through questionnaire.
6. Ability to understand and comply all procedures of the study, and provide written consent.

Exclusion Criteria:

1. Confirmed diagnosis of pneumonia or other disease by chest X ray which would impact on study evaluations.
2. Must require long-term use of NASIDs, corticosteroids or other immunosuppressive agents.
3. Pregnant female.
4. Subjects are not suitable for the conduct of the study for any other reasons, determined by the investigator. For example, subjects who require to use antibiotics, COVID-19 or influenza antiviral drugs. -

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2023-08-07 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint is the "time to symptom-free for fever" which is the days of the symptom-free for fever based on the diary record. | 5 days

SECONDARY OUTCOMES:
the "time to symptom-free for sore throat" will be analyzed as the analysis of the primary efficacy endpoint. | 1 week

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Linkou Chang-Gung Memorial Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-06-27): https://cdn.clinicaltrials.gov/large-docs/93/NCT06086093/Prot_000.pdf